CLINICAL TRIAL: NCT05105906
Title: Post-operative Delirium (POD) Assessment in Patients Undergoing Hip Fracture Surgery
Brief Title: Post-operative Delirium (POD) in Patients Undergoing Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Giuliano Ferrone, M.D., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: FPG ID 3993
Record Dates: First submitted 2021-09-29; First posted 2021-11-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Delirium; Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cognitive tests performed — cognitive tests performed

SUMMARY:
The primary endpoint of the study is the appearance of Post Operative Delirium within the first 3 months.

The secondary endpoints are the development of POCD, dementia of any type of new onset at 12 months, mortality at 30 days, postoperative hospitalization time (including rehabilitation performed within the Polyclinic).. The analysis of the risk factors of POD and their correlation with the development of POCD/Dementia in the post-surgery period will provide important information for the optimization of the management path of these patients at an individual level , with inevitable repercussions on the possibility of reintegration into social and family life

ELIGIBILITY:
Inclusion Criteria:

* Age > 65
* Clinical - radiological presence of hip fracture

Exclusion Criteria:

* Age <65

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All men and women over the age of 65 with clinical-radiological hip fracture presence will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Appearance of POD within the first 3 months | 3 months assessment
  Appearance of Post Operative Delirium within the first 3 months after hip surgery

SECONDARY OUTCOMES:
Development of POCD, dementia of any type of new onset at 12 months, mortality at 30 days, postoperative hospitalization time | 12 months assessment
  Development of Post Operative Cognitive Dysfunction, dementia of any type of new onset at 12 months, mortality at 30 days, postoperative hospitalization time

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Ferrone, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No